CLINICAL TRIAL: NCT05758688
Title: Adjuvant Proton Whole Pelvis Radiation Therapy for Treatment of Post-Surgical Gynecologic Cancers
Brief Title: PROton Therapy for Post Surgical Treatment of GYNecologic Cancer
Acronym: PROPS GYN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 27822; 852760 (Other: University of Pennsylvania)
Record Dates: First submitted 2023-01-24; First posted 2023-03-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer; Uterine Cancer; Endometrial Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Adjuvant Whole Pelvis (WP) Pencil Beam Scanning Proton Radiation (PBS PRT) (Experimental): The study intervention is Whole Pelvis (WP) Pencil Beam Scanning Proton Radiation (PBS PRT) as part of the definitive treatment of gynecologic cancers in the post-hysterectomy, adjuvant setting. Patients will be treated with doses of 45 or 50.4 Gy in 1.8 Gy daily fractions. The volume treated will include the whole pelvis according to Radiation Therapy Oncology Group post-hysterectomy pelvis guidelines.
  Interventions: Radiation: Whole Pelvis (WP) Pencil Beam Scanning Proton Radiation (PBS PRT)

INTERVENTIONS:
Radiation: Whole Pelvis (WP) Pencil Beam Scanning Proton Radiation (PBS PRT) — The study intervention is Whole Pelvis (WP) Pencil Beam Scanning Proton Radiation (PBS PRT) as part of the definitive treatment of gynecologic cancers in the post-hysterectomy, adjuvant setting. Patients will be treated with doses of 45 or 50.4 Gy in 1.8 Gy daily fractions. The volume treated will include the whole pelvis according to Radiation Therapy Oncology Group post-hysterectomy pelvis guidelines.

SUMMARY:
This is a single institution, multi-center, Phase II, single-arm study, using Whole Pelvis (WP) Pencil Beam Scanning Proton Radiation (PBS PRT) in the post-surgical, adjuvant setting for definitive treatment of gynecologic cancers. The purpose of this study is to estimate rate of acute clinician-reported gastrointestinal (GI) toxicity using WP PBS PRT in the definitive treatment of gynecologic cancers in the post-surgical, adjuvant setting.

DETAILED DESCRIPTION:
This is a single institution, multi-site study, and thus will include patients from geographic locations with Penn proton centers in the Philadelphia, Lancaster and South New Jersey area. The study will be conducted at the University of Pennsylvania Department of Radiation Oncology and associated Clinical facilities.

The study intervention is Whole Pelvis (WP) Pencil Beam Scanning Proton Radiation (PBS PRT) as part of the definitive treatment of gynecologic cancers in the post-hysterectomy, adjuvant setting. Patients will be treated with doses of 45 or 50.4 Gy in 1.8 Gy daily fractions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervical or endometrial cancer
* Indication for adjuvant whole pelvic radiation therapy, with or without systemic therapy
* Age of 18 years or older
* Written informed consent
* ECOG of 0-2 within 3 months of enrolling

Exclusion Criteria:

* Prior course of pelvic radiation
* Metastatic disease outside of the pelvis
* Active inflammatory bowel disease
* Incapacity to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Acute clinician-reported gastrointestinal (GI) toxicity. | Up to 6 months after end of treatment at follow up visits
  Determine the rate of acute clinician-reported gastrointestinal (GI), with the Common Terminology Criteria for Adverse Events (CTCAE v5.0) criteria. Acute GI grade 2 or higher toxicity is the primary powering endpoint.

SECONDARY OUTCOMES:
Acute clinician-reported genitourinary (GU) toxicity. | Up to 6 months after end of treatment at follow up visits
  Determine the rate of the acute clinician-reported genitourinary (GU) toxicity, with the Common Terminology Criteria for Adverse Events (CTCAE v5.0) criteria.
Acute patient-reported gastrointestinal (GI) and genitourinary (GU) toxicity and quality of life. | Up to 6 months after end of treatment at follow up visits
  Determine the rate of acute patient-reported gastrointestinal (GI) and genitourinary (GU) toxicity and quality of life using the EPIC urinary and bowel score (expanded prostate cancer index composite) and FACT-Cx.
Loco-regional recurrence free survival, disease free survival, and overall survival. | Up to 2 years
  Determine loco-regional recurrence free survival, disease free survival, and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Neil K Taunk, MD, MSCTS, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Virtua Health, Voorhees Township, New Jersey
  - Lancaster General Health - Ann B. Barshinger Cancer Institute, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania